CLINICAL TRIAL: NCT01532427
Title: ALFApump System Post Marketing Surveillance Registry, In Support of the Following Indication: Automated Removal of Excess Peritoneal Fluid Into the Urinary Bladder in Patients With Cirrhosis or Malignancy, With Persistent or Refractory Ascites
Brief Title: ALFApump System Post Marketing Surveillance Registry
Acronym: 2011-AAR-004
Status: Completed | Type: Observational
Sponsor: Sequana Medical N.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011-AAR-004
Record Dates: First submitted 2012-02-09; First posted 2012-02-14 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Liver Cirrhosis; Refractory Ascites; Malignant Ascites
MeSH Terms: conditions — Liver Cirrhosis; Ascites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a post market surveillance registry to monitor the safety and performance of the ALFApump system.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or recurrent ascites and liver cirrhosis or malignancy
* written informed consent

Exclusion Criteria:

* < 18 years
* pregnant
* not able to use the Smart charger

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Registry will include 200 patients implanted after market approval at up to 25 centres, in patients with liver cirrhosis or malignancy, with persistent or refractory ascites.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Safety | 24 months
  To monitor the safety of the ALFApump System

SECONDARY OUTCOMES:
clinical performance | 24 months
  To monitor clinical performance of the ALFApump System
clinical impact | 24 months
  To monitor the clinical impact of the ALFApump System
usability | 1 month
  To assess the usability of the ALFApump System

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Gottardi, Privatdozent, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (13):
- Germany (8):
  - Uniklinik Dresden, Dresden
  - Klinikum der Johann Wolfgang Goethe Universität, Frankfurt
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Universitätsklinikum Jena, Jena
  - St Georg Klinik, Leipzig
  - Universitätsklinikum Leipzig, AöR, Leipzig
  - Medizinische Klinik, Universitätsmedizin Mannheim, Mannheim
  - Uniklinik Würzburg, Würzburg
- Hosptial Universitari Vall d'Hebron, Barcelona, Spain
- Switzerland (2):
  - Inselspital, Bern
  - University Clinic of Geneva (HUG), Geneva
- United Kingdom (2):
  - The London Clinic, The liver centre, London
  - Freeman Hospital Newcastle on Tyne, Newcastle upon Tyne

REFERENCES:
- [Derived] Stirnimann G, Berg T, Spahr L, Zeuzem S, McPherson S, Lammert F, Storni F, Banz V, Babatz J, Vargas V, Geier A, Engelmann C, Herber A, Trepte C, Capel J, De Gottardi A. Final safety and efficacy results from a 106 real-world patients registry with an ascites-mobilizing pump. Liver Int. 2022 Oct;42(10):2247-2259. doi: 10.1111/liv.15337. Epub 2022 Jul 25. PMID 35686702
- [Derived] Stirnimann G, Berg T, Spahr L, Zeuzem S, McPherson S, Lammert F, Storni F, Banz V, Babatz J, Vargas V, Geier A, Stallmach A, Engelmann C, Trepte C, Capel J, De Gottardi A. Treatment of refractory ascites with an automated low-flow ascites pump in patients with cirrhosis. Aliment Pharmacol Ther. 2017 Nov;46(10):981-991. doi: 10.1111/apt.14331. Epub 2017 Sep 21. PMID 28940225